CLINICAL TRIAL: NCT06098508
Title: The Effects of Osteopathic Manual Treatment on Hemiplegic Shoulder Pain and Upper Extremity Function in Stroke Patients: A Pilot Study
Brief Title: Osteopathic Manual Treatment for Hemiplegic Shoulder Pain and Upper Extremity Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-1051; SMPH/ORTHO&REHAB/REHAB MED (Other: UW Madison); Protocol version 8/8/25 (Other: UW Madison); A536120 (Other: UW Madison)
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Hemiplegic Shoulder Pain; Osteopathic Manipulative Treatment
Keywords: stroke; hemiplegic shoulder pain; Osteopathic Manual Treatment; OMT
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Other members of the study team, such as those who recruit, screen, and coordinate research visits, will be masked. Additionally, the occupational therapist who performs baseline pain ratings and arm function assessments will also be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manual Treatment (Experimental)
  Interventions: Other: Osteopathic Manual Treatment
- Sham Treatment Arm (Sham Comparator)
  Interventions: Other: Sham Treatment

INTERVENTIONS:
Other: Osteopathic Manual Treatment — This study will be using osteopathic manual therapy as the primary intervention. Osteopathic manual therapy (OMT) is a hands-on treatment that is performed by a specially trained physician known as a Doctor of Osteopathic Medicine (DO). This treatment can be used to diagnose and treat somatic dysfunctions, which are palpable areas of tightness, misalignment, and/or restricted motion within the musculoskeletal system and its related vascular and neural structures. A combination of myofascial release, strain/counterstain, soft tissue, balanced ligamentous release, facilitated positional release and muscle energy techniques will be used for the OMT treatment.
  Arms: Osteopathic Manual Treatment
Other: Sham Treatment — The sham treatment will include a hands-on evaluation typically used to diagnose somatic dysfunctions, but no treatment will be performed. The sham treatment will assess the upper extremities/scapulae, ribs, cervical spine, thoracic spine, thoracic inlet, and occipital-atlantal regions.
  Arms: Sham Treatment Arm

SUMMARY:
This study assesses the feasibility and safety of performing osteopathic manual treatment (OMT) for hemiplegic shoulder pain in stroke patients. This study's participants will be adults with a first-time stroke diagnosis in the past 5 years and shoulder pain on the same side affected by stroke. Eligible participants will be placed on study for approximately 6 weeks and given either OMT or a sham treatment each week.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years or older to participate in the study
* Presence of shoulder pain on the side of the body affected by stroke
* Patients must have a diagnosis of a first-time stroke within the past 5 years
* Stroke type must be subcortical, brainstem, and/or right-MCA stroke. Participants with multiple stroke types within the first-time diagnosis may be included

Exclusion Criteria:

* Presence of an active systemic or localized infection requiring antibiotic therapy
* Presence of fracture in the area being treated
* Presence of open wound in the area being treated
* Presence of rheumatoid arthritis
* Presence of known active malignancy
* Presence of shoulder pain on the affected side within 3 months prior to stroke
* Patients with left-MCA stroke diagnosis who demonstrate the presence of aphasia based on the Mississippi Aphasia Screening Test (MAST)
* Patients who demonstrate hemispatial visual neglect based on screening motor-free visual perception test (MFVPT)
* Patients already receiving any type of manual therapy by a certified therapist through their standard-of-care treatment
* Patients who do not wish to participate
* Patients who are not fit as judged by the study team
* Patients who lack the capacity to consent for enrollment in the study based on the University of California San Diego Brief Assessment of Capacity to Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Feasibility Assessment | From enrollment to the end of treatment at 6 weeks
  The study team will assess feasibility by tracking participant recruitment, randomization, and retention. The ability to carry out the intervention protocol to completion in these participants will be assessed. Feasibility will be confirmed if 10 patients are randomized and at least 80% complete the study within the planned 1-year timeline.

SECONDARY OUTCOMES:
Safety Assessment | From enrollment to the end of treatment at 6 weeks
  The study team will also assess the safety of performing osteopathic manual therapy in stroke patients with hemiplegic shoulder pain. Any reported adverse events (AE) and severe adverse events (SAE) will be tracked and monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Mohan, DO, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Health University Ave Rehabilitation Clinic, Middleton, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Preliminary data that has been anonymized may be shared within the academic intuition for research purposes. Once published, data will be shared with the general public. Any data that is published or presented will not be identifiable.
  All data collected during the study will be banked indefinitely after study completion for future research. All participant identifiers will be removed prior to banking the data. The principal investigator and co-investigators of this current study will have access to the stored data. If there is a request for this data to be shared outside of this study team, the PI will decide if the data can be shared and the data will be fully anonymized. This data would be shared for future research related to osteopathic manual therapy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Researchers interested in pursuing OMT research may contact Ashley Mohan, DO, at mohan@rehab.wisc.edu for access to IPD documents.